CLINICAL TRIAL: NCT02792452
Title: Clinical Value of Stress Echocardiography in Moderate Aortic Stenosis
Status: Completed | Type: Observational
Sponsor: London North West Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: AV AS-01
Record Dates: First submitted 2016-05-19; First posted 2016-06-07 (Estimated); Last update posted 2020-02-12 (Actual); Status verified 2020-01

CONDITIONS: Aortic Valve Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The management of symptomatic patients with moderate Aortic Stenosis (AS) remains challenging and tests that would give more definitive answers are needed. The value of increase in Aortic Valve mean Gradient (AVMG), lack of change in Aortic Valve area (AVA) and calculation of valve compliance/resistance during stress echo (SE) in the symptomatic moderate AS population prognostication has to the investigators knowledge not been examined before. Similarly the additive value of myocardial blood flow reserve (MBFR), Computed Tomography (CT) calcium score, speckle tracking echocardiography, carotid ultrasonography, and N-Terminal pro B- type natriuretic peptide B (NT-proBNP) in the prognostication of this population group especially in combination with SE remains unclear.

DETAILED DESCRIPTION:
The prevalence of aortic valve stenosis (AS) has increased over the last few decades due to improvement in life expectancy and a growing elderly population. A wealth of data is available on patients with severe AS, whereas the risk stratification and management of patients with symptomatic moderate AS remains contentious.

Stress echocardiography (SE) is a recognised tool for the risk stratification of patients with asymptomatic severe AS. Exercise is the preferred mode of stress in this group, as it provides important prognostic information- such as presence of symptoms, overall exercise capacity and precipitation of hypotension. Significant increase in mean gradient (MG) (MG >20mmHg) is an independent predictor of valve intervention or cardiovascular death, similar to older age, diabetes and high resting gradient and this is recognised in international guidelines as a parameter to risk stratify asymptomatic severe AS. The increase in MG in the context of increasing transvalvular flow during exercise is usually accompanied by little or no change in aortic valve area (AVA). Thus, mechanistically, the increase in MG is associated with worse outcome because it reflects the intrinsic non-compliance of the aortic valve and hence resistance. A compliant valve will open to accommodate the increased flow during stress, whereas a fixed valve orifice will not, resulting in increased gradients. It is therefore advised that these patients with asymptomatic severe AS and significant increase in MG during exercise may be reasonably considered for aortic valve intervention.

In moderate AS current guidelines recommend Aortic Valve replacement (AVR) only when other cardiac surgery (coronary artery bypass grafting) is planned (class IIa). This is because patients with moderate AS are a heterogeneous group with regard to the risk of adverse events: some have indeed rapid progression to severe AS, and/or Left Ventricular (LV) dysfunction and cardiovascular death, whereas others remain stable for many years. Overall moderate AS carries a substantial risk of death or valve intervention, with the estimated likelihood of event free survival at 4 years being 55-60%. Furthermore the presence of symptoms increases the overall likelihood of risk in moderate AS, as there is a significant difference in outcome between minimally symptomatic and symptomatic moderate AS. It maybe hypothesised that patients with moderate AS and symptoms in the absence of myocardial ischaemia due to flow-limiting coronary artery disease likely has the same valve hemodynamics as one with severe AS, particularly decreased valve compliance/increased resistance. These characteristics are likely to manifest during exercise when transvalvular flow is increased resulting in significant increase in gradient with little change in AVA. Accordingly, resting AVA and MG may not be the best parameters for determining suitability for valve intervention, particularly as the overall mortality of symptomatic moderate aortic stenosis approaches that of symptomatic severe AS. However, clear criteria that risk-stratify patients with symptomatic moderate AS and guide timing for intervention do not currently exist.

Accordingly the role of SE could be expanded beyond assessment of risk in asymptomatic severe AS to improve risk stratification in patients with symptomatic moderate AS. This is on the assumption that moderate AS associated with symptoms of breathlessness, chest pain or syncope is likely to have the same characteristics as severe AS. This means that during SE in moderate symptomatic AS one would expect the AVA to remain unchanged, the valve resistance to be elevated and the MG to increase.

Furthermore during SE apart from valve related indices that determine severity (AVA, MG), myocardial blood flow reserve (MBFR) has been shown to correlate with severity of AS; reduced MBFR is seen in severe AS whereas MBFR<1.8 has an accuracy of 85% for distinguishing severe from non-severe AS. It could therefore be that MBFR can also contribute in the risk stratification of symptomatic moderate AS.

It has been suggested that several other tests could contribute to the risk stratification of AS i.e. CT calcium score, speckle tracking echocardiography, carotid ultrasonography, and N-terminal pro-brain natriuretic peptide (NT-proBNP). Specifically it has been shown that aortic valve calcium score correlates with AS severity and that there is moderate agreement between AVA as defined by American College of Cardiology (ACC) guidelines and the degree of AS determined from AV calcium score. Basal and global longitudinal strain (GLS) have been found to be independently associated both with the severity of AS and the presence of symptoms. Furthermore GLS can predict all-cause mortality in patients with AS and could therefore improve the identification of the optimal timing for AV replacement. The severity of AS in general has also been shown to correspond to an increase of carotid plaque and intima media thickness (IMT). Finally NT-proBNP values correlate with the severity of AS and in moderate AS, NT-proBNP can differentiate between symptomatic and asymptomatic status.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Moderate AS with AVA between 1-1.4cm2, and AVMG<40 millimetres of Mercury (mmHg); and
* Left Ventricular Ejection Fraction (LVEF) ≥50%; and
* Cardiac related symptoms; shortness of breath, chest pain or syncope.

Exclusion Criteria:

* Inability to exercise and undertake pharmacological stress, ie previously known intolerance to dobutamine;
* Severe aortic or mitral regurgitation or severe mitral stenosis;
* Significant pulmonary disease like severe (Chronic Obstructive Pulmonary Disease (COPD) or pulmonary fibrosis;
* Atrial fibrillation;
* Inability to provide informed consent;
* Pregnancy;
* Other known non-cardiovascular disease associated with poor prognosis like metastatic cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Suitable patients with moderate Aortic stenosis will be identified from the Echocardiography labs of the two trusts (London North West Healthcare NHS Trust and Royal Brompton Hospital) and will be approached for enrolment in the study.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2016-09; Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Death (cardiovascular/all cause) | between baseline and two years
Hospitalisation for heart failure | between baseline and two years
Aortic valve replacement (TAVI or surgical AVR) | between baseline and two years

SECONDARY OUTCOMES:
Change in AS severity (progression to severe) as measured by quantitive echocardiography | Between baseline and one year
change in LV systolic function as measured by quantitive echocardiography | Between baseline and one year

CONTACTS AND LOCATIONS:
Overall Officials: Roxy Senior, MD,DM,FRCP, Study Director — London North West Healthcare NHS Trust
Locations (1):
- Northwick Park Hospital, Harrow, MIddx, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Patient scan results will be shared with their referring physician